CLINICAL TRIAL: NCT06279494
Title: Sirolimus+Abatacept+Mycophenolate Mofetil Regimen for Prophylaxis of Acute Graft-versus-host Disease (aGvHD) in Patients Receiving Haploidentical Hematopoietic Stem Cell Transplantation (Haplo-HSCT) Who Are Intolerant to Calcineurin Inhibitor
Brief Title: Sirolimus+Abatacept+Mycophenolate Mofetil for Prophylaxis of aGVHD in Patients Receiving Haplo-HSCT Who Are Intolerant to Calcineurin Inhibitors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Prof., Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Sirolimus for GVHD prophylaxis
Record Dates: First submitted 2024-02-09; First posted 2024-02-28 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Acute Leukemia; Myelodysplastic Syndromes; Severe Aplastic Anemia
Keywords: Abatacept; Mycophenolate Mofetil; Sirolimus; Graft-versus-host-disease; Haploidentical; Calcineurin Inhibitor
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia, Aplastic; Graft vs Host Disease | interventions — Sirolimus; Abatacept

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sirolimus+Abatacept+Mycophenolate mofetil (MMF)+anti-thymocyte globulin (ATG) (Experimental): Patients receiving haplo-HSCT who are intolerant to calcineurin inhibitors would receive Sirolimus+Abatacept+MMF+ATG (SAMA) for prophylaxis of aGVHD
  Interventions: Drug: Sirolimus; Drug: Abatacept; Drug: MMF; Drug: ATG

INTERVENTIONS:
Drug: Sirolimus — Orally (concentration 5-10ng/ml) from -1 to +100d post haplo-HSCT
Drug: Abatacept — 5mg/kg subcutaneous, -1/+5/+14/+28/+42/+56d post haplo-HSCT
Drug: MMF — 0.5g bid orally, from -3d to +60d post haplo-HSCT
Drug: ATG — 2.5 mg/kg, from -5d to -2d

SUMMARY:
Graft-versus-host disease (GVHD) is an important complication after transplantation, with an incidence of 40-60%, which can increase non-relapse mortality if poorly controlled. At present, the standard prophylaxis for GVHD is cyclosporine combined with methotrexate. However, calcineurin inhibitors (CNI) can cause some vital side effects, which are not tolerated by some patients. Therefore, this study aims to explore the safety and efficacy of Sirolimus in combination with Abatacept and Mycophenolate Mofetil for the prophylaxis of GVHD in patients with haplo-HSCT who are intolerant to calcineurin inhibitors.

ELIGIBILITY:
Inclusion criteria:

1. Primary disease: hematological malignancies (including acute leukemia, myelodysplastic syndromes), nonmalignant disorders (including severe aplastic anaemia)
2. Contraindication or intolerance to CNI

   1. Glomerular filtration rate (GFR) 60-89 ml/min/1.73m2 before transplantation or allergy to CNI
   2. Intolerance to CNI during conditioning or within +45 days post transplantation, such as CNI nephrotoxicity (creatinine higher than the upper limit of normal), uncontrolled hypertension, neurological toxicity, or other conditions deemed by physician to be inappropriate for CNI
3. Receiving haplo-HSCT for the first time

Exclusion Criteria:

1. Allergy or intolerance to study drugs
2. Active infection
3. Active GVHD
4. Transplantation-associated thrombotic microangiopathy
5. Key organ dysfunction: liver injury (total bilirubin more than 2 upper limit of normal) or heart injury (symptomatic heart failure or ejection fraction<50%)
6. Eastern Cooperative Oncology Group (ECOG) score >2
7. Expected survival time <30 days
8. Patients could not cooperate

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Grade 2-4 aGVHD within 100 days post transplantation | Participants will be followed for an expected average of 100 days post transplantation

SECONDARY OUTCOMES:
Incidence of chronic GVHD (cGVHD) within 1 year post transplantation | Participants will be followed for an expected average of 1 year
Incidence of thrombotic microangiopathy within 1 year post transplantation | Participants will be followed for an expected average of 1 year

OTHER OUTCOMES:
Cumulative incidence of relapse | Participants will be followed for an expected average of 1 year
Transplant-related mortality | Participants will be followed for an expected average of 1 year
Overall survival | Participants will be followed for an expected average of 1 year
Incidence of cytomegalovirus (CMV) and Epstein-Barr virus (EBV) | Participants will be followed for an expected average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Jun Huang, Principal Investigator — Institute of Hematology, Peking University